# <u>Title: The prevalence and association of anxiety and sleep disturbances among medical students: A cross-sectional study</u>

## Recent updated Date: April 29,2025

It is a cross-sectional study conducted in December 2024 with the consent of 200 undergraduate medical students of a tertiary care hospital affiliated medical college, who qualified as per the inclusion criteria.

#### Inclusion criteria:

• All the students of MBBS Phase-II.

#### Exclusion criteria:

- Students with prior diagnosed Sleep disorders
- Students with prior diagnosed co-morbidities
- Students unable/unwilling to answer the question.

### **Statistical analysis:**

The qualitative data on the Categorical variables will be presented in terms of numbers and extended in percentages (%). The following statistical tests were applied to the results:

- 1. In the analysis of this study, the Chi-Square test will be used to test the significance of the difference between the groups of the study about the Qualitative variables.
- 2. This will be rated based on the degree of statistical significance, whereby a p-value < 0.05 will be taken, otherwise, the given value will be regarded as statistically significant.

The data entry will be done in the Microsoft Excel spreadsheet, and the final analysis will be done using Statistical Package for Social Sciences (SPSS) software, IBM, Chicago, USA, version 25.0.

Note: Informed Consent Forms are not being shared here publicly to maintain participant confidentiality.